CLINICAL TRIAL: NCT00993889
Title: Virtual Reality Analgesia During Pediatric Physical Therapy
Acronym: VRD/Peds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, David R. Patterson, PhD.ABPP. Professor, National Institute of General Medical Sciences (NIGMS)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 36154-C
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Burn
Keywords: Virtual Reality Peds
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- VR during Physical Therapy (Experimental): The subject will receive virtual reality during painful physical therapy sessions.
  Interventions: Behavioral: VR during Physical Therapy
- VR background pain (Experimental): The subjects receives virtual reality, not during a physical therapy procedure, another time of the day for background pain.
  Interventions: Behavioral: VR Background Pain
- No VR (Experimental): The subject will receive the usual standard treatment. At the end of the study, before being discharged from the hospital, the subject can experience the VR, not during a procedure.
  Interventions: Behavioral: NO VR

INTERVENTIONS:
Behavioral: VR during Physical Therapy — Virtual Reality will be performed during a painful physical therapy procedure.
  Arms: VR during Physical Therapy
Behavioral: VR Background Pain — Virtual Reality is used at anytime during the day for the background pain, not during physical therapy.
  Arms: VR background pain
Behavioral: NO VR — The subject will receive the usual standard treatment. At the end of the study, before being discharged from the hospital, the subject can experience the VR, not during a procedure.
  Arms: No VR

SUMMARY:
We would like to determine whether Virtual Reality (VR) analgesia continues to be effective for reducing pain when administered for a clinically relevant treatment duration over multiple, repeated exposures (i.e., up to ten sessions of physical therapy per patient).

DETAILED DESCRIPTION:
This study is done in a hospital for inpatients pediatrics. By randomization some subjects will immersive Virtual Reality (VR) during a painful procedure on daily basis up to 10 days to see whether this will reduce the pain and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 8 years up to 20 yrs old
* Compliant and able to complete subject evaluation
* A minimum of 3 days of physical therapy, one physical therapy session per day
* No history of psychiatric (DSM-IV-R Axis I) or developmental disorder that would interfere with decisional capacity
* Not demonstrating delirium, psychosis, or any form of Organic Brain Disorder that would interfere with decisional capacity
* Able to communicate verbally
* Able to take oral medications
* English-speaking

Exclusion Criteria:

* - Age less than 8 years, or greater than 20 years.
* Not capable of indicating pain intensity
* Not capable of filling out study measures
* Hospitalization of fewer than 3 days
* Evidence of traumatic brain injury
* History of psychiatric (DSM-IV-R Axis I) disorder as evidenced in the admitting RN and MD admission notes, if interfering with decisional capacity
* Demonstrating delirium, psychosis or any form of Organic Brain Disorder and associated memory problems that would interfere with decisional capacity
* Unable to communicate verbally
* Unable to take oral medications
* History of sig. cardiac, endocrine, neurologic, metabolic, respiratory, gastrointestinal or genitourinary impairment that would interfere with treatment or decisional capacity
* Receiving prophylaxis for alcohol or drug withdrawal
* Developmental disability that would interfere with decisional capacity
* Face/head/neck injuries preventing helmet use
* Non-English-speaking
* Extreme susceptibility to motion sickness
* Seizure history

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2009-05; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Pain and anxiety | pre and post procedure

CONTACTS AND LOCATIONS:
Overall Officials: David R Patterson, Ph.D., Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States